CLINICAL TRIAL: NCT06279962
Title: Measuring Level of Mental Illness Stigma Based on Condition and Gender
Brief Title: Survey Experiment to Estimate Level of Mental Illness Stigma Based on Condition and Gender
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Empower Through Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2000034605_a
Record Dates: First submitted 2024-02-14; First posted 2024-02-28 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Mental Illness; Stigma, Social
Keywords: stigma; mental illness; low-income country
MeSH Terms: conditions — Mental Disorders; Social Stigma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Experimental: V1: Woman with Major Depressive Disorder (Experimental): Depicting a young woman with symptomatic major depressive disorder
  Interventions: Other: Survey questionnaire
- Experimental: V2: Man with Major Depressive Disorder (Experimental): Depicting a young man with symptomatic major depressive disorder
  Interventions: Other: Survey questionnaire
- Experimental: V3: Man with Generalized Anxiety Disorder (Experimental): Depicting a young man with symptomatic generalized anxiety disorder
  Interventions: Other: Survey questionnaire
- Experimental: V4: Woman with Generalized Anxiety Disorder (Experimental): Depicting a young woman with symptomatic generalized anxiety disorder
  Interventions: Other: Survey questionnaire
- Experimental: V5: Woman with Schizophrenia (Experimental): Depicting a young woman with symptomatic schizophrenia
  Interventions: Other: Survey questionnaire
- Experimental: V6: Man with Schizophrenia (Experimental): Depicting a young man with symptomatic schizophrenia
  Interventions: Other: Survey questionnaire
- Experimental: V7: Woman with Alcohol Use Disorder (Experimental): Depicting a young woman with symptomatic alcohol use disorder
  Interventions: Other: Survey questionnaire
- Experimental: V8: Man with Alcohol Use Disorder (Experimental): Depicting a young man with symptomatic alcohol use disorder
  Interventions: Other: Survey questionnaire

INTERVENTIONS:
Other: Survey questionnaire — The intervention is being assigned to one of the 8 different versions of the survey vignette.

SUMMARY:
This study aims to measure levels of mental illness stigma based on condition and gender of the participants and individual portrayed with mental illness.

DETAILED DESCRIPTION:
This study aims to measure levels of mental illness stigma based on condition and gender of the participants and individual portrayed with mental illness. This study utilizes eight vignettes portraying different mental illnesses and genders to measure the levels of mental illness stigma in the general community in rural Uganda.

ELIGIBILITY:
Inclusion Criteria:

* All adults who consider Buyende District their primary residence and who are capable of providing consent

Exclusion Criteria:

* Minors younger than 18 years of age
* Persons who do not consider Buyende District their primary place of residence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Level of acceptance for the individual depicted in the vignette as measured by PERSONAL ACCEPTANCE SCALE | Study period. For each interview, approximately 60 minutes.
  The PAS is a 9-item questionnaire targeted to public stigma, the "negative attitudes, beliefs, and behaviors held within a community" against individuals with mental illness. Each yes adds one point to the scale, and five questions from each scale were reverse-scored to match the direction of the scale. The total number of points was divided by the number of questions (nine) and multiplied by ten to generate numbers between zero and ten for comparison purposes to the Broad Acceptance Scale. Higher scores indicated more acceptance and less stigma towards mental illness, while lower scores indicated less acceptance and more stigma towards mental illness.
Level of acceptance for the individual depicted in the vignette as measured by BROAD ACCEPTANCE SCALE | Study period. For each interview, approximately 60 minutes.
  The BAS is a 9-item questionnaire targeted to structural stigma, the "societal-level conditions, cultural norms, and institutional practices that constrain the opportunities, resources, and wellbeing" for individuals with mental illness. Each yes adds one point to the scale, and five questions from each scale were reverse-scored to match the direction of the scale. There were ten questions, therefore it generated a score between zero and ten. Higher scores indicated more acceptance and less stigma towards mental illness, while lower scores indicated less acceptance and more stigma towards mental illness.

CONTACTS AND LOCATIONS:
Locations (1):
- Empowerment to Heal - Uganda, Iganga, Uganda

IPD SHARING:
Plan to Share IPD: Undecided